CLINICAL TRIAL: NCT03842592
Title: Quantification of Ventricular Arrhythmia After Myocarditis in Sportsman
Brief Title: Ventricular Arrhythmia After Myocarditis in Sportsman
Acronym: ARYMYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018-A03328-47
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Myocarditis Acute; Ventricular Arrythmia
MeSH Terms: interventions — Exercise Test; Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- To establish the rhythmic load of sports patients at a distance from a first episode of myocarditis. (Other): Stress testing and 24-hour Holter ECG are the tools currently recommended for assessing rhythmic load and, consequently rhythmic risk. These investigations will be perform at 1 years after myocardite.
  Interventions: Diagnostic Test: Treadmill Stress test

INTERVENTIONS:
Diagnostic Test: Treadmill Stress test — Ventricular arrhythmia will be assessed by ECG Holter and during treadmill stress test, both being performed 3 months and 1 year after acute myocarditis
  Other Names: ECG Holter

SUMMARY:
The study aims to assess the prevalence of ventricular rhythmic disorder after an acute myocarditis in sportsmen.

50 patients with acute myocarditis, confirmed by MRI, will be assessed by ECG Holter and Treadmill stress test during a 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* acute myocarditis, diagnosed on the association of (a) recent viral infection (upper airway, gastro-intestinal) , (b) troponin increase, and (c) chest pain AND myocarditis confirmed by cardiac magnetic resonance 2 out of 3 Lake Louise criteria, either T2 hypersignal, early enhancement or late gadolinium enhancement.
* regular physical activity, recreational or competitive: >=4 hours weekly
* written informed consent

Exclusion Criteria:

* coronary artery disease
* acute inflammatory cardiomyopathy (sarcoidosis, fulminant myocarditis, Tako Tsubo, eosinophilic myocarditis, Lyme disease)
* history of myocarditis
* contra-indication to cardiac MRI
* patient unable to perform a treadmill stress test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Complex ventricular arrhythmia | any timepoint: 3 month and/or 1 year
  any ventricular tachycardia (triplet or more), ventricular fibrillation (observed on ECG Holter or during stress test)

SECONDARY OUTCOMES:
In-hospital ventricular arrhythmia | up to 2 weeks after admission
  any ventricular tachycardia (triplet or more), ventricular fibrillation, recorded on ECG monitoring
Left Ventricular remodeling | between baseline and 3 months
  Change in LV volumes during time
Left ventricular fibrosis | between baseline and 3 months
  Change in interstitial fibrosis by T1 mapping cardiac magnetic resonnance
Major adverse cardio vascular event | up to 2 years after inclusion
  CV death, sudden cardiac death, cardiac graft or haemodynamic support, hospitalisation for heart failure, new event of myocarditis
return to physical activity | up to 2 years after inclusion
  defined as at least 75% of exercising time (in hours per week)

CONTACTS AND LOCATIONS:
Overall Officials: Loïc BIERE, MD PhD, Principal Investigator — Department of Cardiology, University Hospital of Angers (France)
Locations (4):
- France (4):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Lariboisière University Hospital - AP-HP, Paris
  - Rennes University Hospital, Rennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Te ALD, Wu TC, Lin YJ, Chen YY, Chung FP, Chang SL, Lo LW, Hu YF, Tuan TC, Chao TF, Liao JN, Chien KL, Lin CY, Chang YT, Chen SA. Increased risk of ventricular tachycardia and cardiovascular death in patients with myocarditis during the long-term follow-up: A national representative cohort from the National Health Insurance Research Database. Medicine (Baltimore). 2017 May;96(18):e6633. doi: 10.1097/MD.0000000000006633. PMID 28471960
- [Background] Maron BJ, Doerer JJ, Haas TS, Tierney DM, Mueller FO. Sudden deaths in young competitive athletes: analysis of 1866 deaths in the United States, 1980-2006. Circulation. 2009 Mar 3;119(8):1085-92. doi: 10.1161/CIRCULATIONAHA.108.804617. Epub 2009 Feb 16. PMID 19221222
- [Background] Maron BJ, Udelson JE, Bonow RO, Nishimura RA, Ackerman MJ, Estes NA 3rd, Cooper LT Jr, Link MS, Maron MS; American Heart Association Electrocardiography and Arrhythmias Committee of Council on Clinical Cardiology, Council on Cardiovascular Disease in Young, Council on Cardiovascular and Stroke Nursing, Council on Functional Genomics and Translational Biology, and American College of Cardiology. Eligibility and Disqualification Recommendations for Competitive Athletes With Cardiovascular Abnormalities: Task Force 3: Hypertrophic Cardiomyopathy, Arrhythmogenic Right Ventricular Cardiomyopathy and Other Cardiomyopathies, and Myocarditis: A Scientific Statement From the American Heart Association and American College of Cardiology. Circulation. 2015 Dec 1;132(22):e273-80. doi: 10.1161/CIR.0000000000000239. Epub 2015 Nov 2. No abstract available. PMID 26621644
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828